CLINICAL TRIAL: NCT03869216
Title: Fostering Shared Decision-making About Prostate Cancer Screening Among Clinicians and African American Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xavier University of Louisiana. (Other)
Collaborators: Tulane University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB684-20; U54MD007595 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Primary Care; PSA-screening; African American males
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Care Provider
Masking Description: The patients are the unit of randomization and physicians do not know what patients are assigned to the intervention or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention will receive the educational intervention
  Interventions: Behavioral: Educational Shared Decision-Making Intervention
- Usual Care (No Intervention): Patients in the control arm will receive usual care

INTERVENTIONS:
Behavioral: Educational Shared Decision-Making Intervention — The intervention includes a web-based patients' decision aid about PSA-based prostate cancer screening, risks and preferences. The providers receive a summary of the USPSTF 2018 guidelines and main components of the Agency for Healthcare Research and Quality (AHRQ) SHARE curriculum, a link to a video of a prototypical shared decision making conversation, and a laminated shared decision making reminder card.
  Arms: Intervention

SUMMARY:
This behavioral clinical trial assesses the efficacy of a educational intervention to increase shared decision making about prostate-specific antigen (PSA)-based screening for prostate cancer among African American males. Half of participants will receive a multimedia educational intervention, while the other half will receive usual care.

DETAILED DESCRIPTION:
The 2018 U.S. Preventive Services Task Force (USPSTF) final recommendation states that male patients and their providers engage in a shared-decision making process about the benefits and harms of PSA-based screening. As characterized by the USPSTF, these conversations are particularly important for African American men given increased ambiguity due to the lack of PSA-based research specific to this population and increased risk of prostate cancer mortality attributed to late stage at diagnosis and more aggressive prostate cancer phenotypes seen in African American men.

The goal of this randomized behavioral clinical trial is to advance the translation path of implementing the decision-making process in clinical encounters by evaluating the efficacy of an educational intervention for African American males to increase shared decision making about PSA-screening versus usual care. The intervention will use multimedia educational training materials to increase understanding of prostate cancer, PSA-based screening, and shared decision making among patients and their primary care providers (PCPs).

ELIGIBILITY:
Patient Inclusion Criteria:

* Receiving care at the clinical sites
* Identify as African American male
* Ages 40-69 years old

Patient Exclusion Criteria:

* Personal history of prostate cancer at the time of consent
* Cognitive impairment that would interfere with participation in the study
* Unable to complete any aspect of the intervention within the specified time limit

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Echeverri, PhD, MSc, Principal Investigator — Xavier University of Louisiana.
Locations (1):
- Tulane Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified summary of participant data for all primary and secondary outcomes measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access request will be reviewed by the Institutional Review Board (IRB) and principal investigators. Requestors will be required to sign a Data Access Agreement

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective participants were identified through the medical records and were invited to participate in the study. Those willing to participate were enrolled in the study after signing the consent and HIPPA forms. Participants were had the option to opt out of the study anytime.
Pre-assignment Details: After completing the baseline, participants were assigned randomly to the intervention or control arms
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 80 | 81
Completed Baseline | 79 | 76
Completed the Intervention | 73 | 0
Had the Medical Appointment (During the medical appointment patient and physician discuss about risks, benefits and decision to have or not have the Prostate-Specific Antigen (PSA) screening test for prostate cancer) | 62 | 64
Completed Follow-up | 60 | 53
Completed | 60 | 53
Not Completed | 20 | 28
Not completed — prostate removed during the study | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 3 | 12
Not completed — Changed clinical site or moved out of city | 5 | 9
Not completed — No primary care appointment scheduled | 10 | 4
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 79 | 76 | 155
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 10 | 18 | 28
  50-59 years old | 30 | 27 | 57
  60-69 years old | 39 | 31 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 79 | 76 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 79 | 76 | 155
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 79 | 76 | 155
Participants with a family history of prostate cancer [Count of Participants; unit: Participants]
  No family history | 66 | 58 | 124
  Have family history | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision-making
Description: The Observing Patient Involvement (OPTION) Scale was used for the coding of the SDM. The total OPTION scale ranges from 0 to 48. Higher values on the scale mean higher patient involvement in the decision-making process.
Time Frame: One month after audio-recorded visit
Population: The OPTION Scale was applied only to patients who had attended the medical appointment (62 in the intervention group, and 64 in the control group). Because one recording in the control group could not be completed (the audio-recording device was damaged), only 63 recordings were evaluated in that group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 62 | 63
Units on a scale | 12.54 (11.0198) | 12.15 (10.4026)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; H0:muI = muC; Test type: Superiority; p = 0.8388, t-test, 2 sided; Mean Difference (Final Values) = 0.395, 95% CI 2-sided [-3.40 to 4.19], Standard Error of Mean 1.916 — Intervention - Control

2. Secondary Outcome: Quality of Decision (QD)
Description: The total QD score ranges from 0 to 100. Higher percentage scores mean higher quality of the decision made.
Time Frame: Up to 24 weeks after the audio-recorded visit
Population: The QD was assessed only for patients who completed the follow-up (60 in the intervention group, and 53 in the control group).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 60 | 53
units on a scale | 82.23 (13.503) | 80.45 (13.925)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; H0:muI = muC; Test type: Superiority; p = 0.4929, t-test, 2 sided; Mean Difference (Final Values) = 1.781, 95% CI 2-sided [-3.35 to 6.91], Standard Error of Mean 2.588

3. Other Pre Specified Outcome: Acceptability
Description: Participants complete a structured questionnaire to rate the acceptability of the enrollment process, study procedures, and their overall satisfaction with the study. The score ranges from 10 to 50. Higher scores mean higher acceptability of study procedures.
Time Frame: Through study completion, an average of 1 year
Population: Acceptability was assessed only for patients who completed the follow-up (60 in the intervention group, and 53 in the control group).
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 60 | 53
unit on a scale | 42.43 (5.318) | 43.17 (4.590)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; H0:muI = muC; Test type: Superiority — Intervention - Control; p = 0.4312, t-test, 2 sided; Mean Difference (Final Values) = -0.735, 95% CI 2-sided [-2.58 to 1.11], Standard Error of Mean 0.932

4. Secondary Outcome: Preference-Congruent Decision Making
Description: The Intention-to-Screen score ranges from 0 to 1. Score = 0 means no intention to receive the PSA test while score = 1 means intention to receive the PSA test.
  Preference-concordant decision making will be scored as 1 (POSITIVE) for those patients with Intention-to-Screen value = 1 who actually receive the PSA test during the study timeframe, or for those patients with Intention-to-Screen value = 0 who did not receive it.
  Preference-concordant decision making will be scored as 0 (NEGATIVE) for those patients with Intention-to-Screen value = 1 who did not receive the PSA test during the study timeframe, or for those patients with Intention-to-Screen value = 0 who did receive it.
  A congruence score of 1 means congruence between patient intention and real action, while a congruence score of 0 means patient in congruence between intention and real action.
Time Frame: Through study completion, an average of 1 year
Population: Congruence was assessed only for patients who completed the follow-up (60 in the intervention group, and 53 in the control group).
Measure: Number; unit: Number of participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 60 | 53
Number of participants
  Participants with Congruence Score = 1 | 36 | 40
  Participants with Congruence Score = 0 | 24 | 13
Statistical Analysis 1: Comparison: Intervention vs Usual Care; H0: piI = piC; Test type: Superiority; p = 0.1216, t-test, 2 sided; Chi Square Test gives same results; Difference in Proportions = -0.1548, 95% CI 2-sided [-0.342 to 0.033], Standard Error of Mean 0.087 — Intervention - Control

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 12 months
Description: This is an educational intervention that did not cause any risk to participants for serious adverse events. During the follow-up call, we recorded information about participants' life events such as being diagnosed with prostate cancer or passing away for natural causes, although these events were not directly related to their participation in the study.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/79 | 1/76
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/76
Other Adverse Events (participants affected / at risk) | 0/79 | 0/76

LIMITATIONS AND CAVEATS:
Significant delays in the advance of the study, were caused by events that were not under our control: Coronavirus disease (COVID19) pandemic and major Hurricanes Zeta and Ida). Because of the restrictions in the city and clinics, several participants moved out and/or did not update their contact information. To address COVID19 restrictions it was necessary to update the study protocol to conduct all activities online and have the new Institutional Review Board approvals in the clinical sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03869216/Prot_000.pdf